CLINICAL TRIAL: NCT00436384
Title: Cell Mediated Immunity and the Prediction of CMV Infection In Solid Organ Transplant Recipients
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Other Study IDs: 05-0265-AE
Record Dates: First submitted 2007-02-15; First posted 2007-02-19 (Estimated); Last update posted 2008-04-16 (Estimated); Status verified 2007-02

CONDITIONS: Transplant
Keywords: liver transplant; lung transplant; kidney transplant; heart transplant; CMV CMI

INTERVENTIONS:
Procedure: Monitoring-blood samples drawn for CMV testing

SUMMARY:
Cytomegalovirus (CMV) is a common cause of illness in patients who have undergone a transplant. Serious infections due to CMV can affect many parts of the body including the lungs, the gut, and the liver. Since transplant recipients are at risk for CMV or have evidence of infection with CMV, they are given an antiviral drug (usually ganciclovir or valganciclovir). Despite this, there are a chance that CMV infection may cause problems in the future. The purpose of this study is to assess how well patients'immune systems responds to the CMV virus, so that in the future it may be possible to predict which patients are at highest risk of CMV.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients who fulfill the following criteria are eligible for inclusion.

  * CMV D+/R- liver, kidney and heart recipient
  * CMV R+ liver,kidney and heart recipients who have received thymoglobulin induction therapy.
  * D+/R- and R+ lung transplant recipients.
  * Able to give written informed consent
  * Are willing and able to comply with the protocol
  * Age >=18 years

Exclusion Criteria:

* Patient unwilling or unable to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2005-11; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Atul Humar, MD, Principal Investigator — University Health Network, Toronto; Deepali Kumar, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada